CLINICAL TRIAL: NCT05951192
Title: A Prospective Interventional Study Assessing the Clinical and Operational Effectiveness of Transitioning From Mircera to Daprodustat for the Treatment of Anemia in End Stage Kidney Disease
Acronym: ROQ-IT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: USRC Kidney Research (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USRC-2023-001
Record Dates: First submitted 2023-06-02; First posted 2023-07-18 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Anemia; Renal Insufficiency, Chronic; Renal Anemia
Keywords: daprodustat; mircera
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Commercial daprodustat (Experimental): Prescription of oral daprodustat in accordance with the FDA approved package label.
  Interventions: Drug: Daprodustat

INTERVENTIONS:
Drug: Daprodustat — Commercially manufactured daprodustat (JESDUVROQ) is provided in tablet strengths of 1, 2, 4, 6 and 8 mg. Tablets will be taken whole and patients will be instructed not to cut, crush, or chew tablets.
  Other Names: JESDUVROQ

SUMMARY:
Investigator-initiated, interventional, prospective study to assess the clinical and operational effectiveness of daprodustat in adult patients receiving in center hemodialysis or peritoneal home dialysis who are transitioning from Mircera to daprodustat.

DETAILED DESCRIPTION:
Investigator-initiated, multicenter, prospective, interventional study to determine the clinical and operational effectiveness of transitioning from intravenous or subcutaneous Mircera to oral daily daprodustat as assessed by change in hemoglobin. This trial will be conducted at up to 40 United States Renal Care sites in the United States and will enroll approximately 200 patients (~150 in-center hemodialysis and ~50 home dialysis patients).

Participants who are prescribed daprodustat by their treating physician and have taken at least a single dose of daprodustat will be considered enrolled into the clinical trial. After the prescription of daprodustat by the treating physician, each subject will be followed prospectively for a treatment period of approximately 120 days.

Subjects taking daprodustat will not have any in-person study related visits and will follow their usual schedule with regard to standard of care. Standard of care laboratory assessments as ordered by the primary nephrologist will be utilized. Twice monthly hemoglobin collection and monitoring will be required as part of the standard of care laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥18 years old.
2. Diagnosis of end stage kidney disease and receiving maintenance dialysis (in-center hemodialysis or peritoneal dialysis) for ≥ 4 months.
3. Has received at least a single dose of Mircera within 45 days prior to prescription of Daprodustat by treating physician.
4. Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure.

Exclusion Criteria:

1. A known allergy or intolerance to daprodustat or any of its constituents.
2. Uncontrolled hypertension.
3. Active malignancy as documented in electronic medical record.
4. Concomitant use of a strong CYP2C8 inhibitor such as gemfibrozil.
5. Severe hepatic impairment as documented in the electronic medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin from baseline to the effectiveness evaluation period | 120 days
  Change in hemoglobin from baseline (defined as the mean of all available hemoglobin values obtained in the 30 days prior to Day 1) to the effectiveness evaluation period (mean of all available hemoglobin values obtained in the 30 days prior to Day 120).

SECONDARY OUTCOMES:
The number/proportion of subjects with a hemoglobin in target range of 10-11 g/dL from baseline to effectiveness evaluation period | 120 days
  The number/proportion of subjects with a hemoglobin in target range of 10-11 g/dL from baseline to effectiveness evaluation period
The number/proportion of subjects with a change in hemoglobin under 0.5 g/dL from baseline to effectiveness evaluation period | 120 days
  The number/proportion of subjects with a change in hemoglobin under 0.5 g/dL from baseline to effectiveness evaluation period
Number of hemoglobin excursions that are < 8.5 g/dL or ≥ 12 g/dL during the treatment period. | 120 days
  Number of hemoglobin excursions that are < 8.5 g/dL or ≥ 12 g/dL during the treatment period.
Number of dose adjustments in daprodustat per patient during the treatment period | 120 days
  Number of dose adjustments in daprodustat per patient during the treatment period
Number of subjects retained on daprodustat therapy from Day 1 through Day 120 | 120 days
  Number of subjects retained on daprodustat therapy from Day 1 through Day 120
The number/proportion of subjects who receive a refill prescription with the correct prescribed dose with no gap (0 days) in drug supply from the previous prescription | 120 days
  The number/proportion of subjects who receive a refill prescription with the correct prescribed dose with no gap (0 days) in drug supply from the previous prescription
The time (in days) from initial and refill prescription to delivery to patient | 120 days
  The time (in days) from initial and refill prescription to delivery to patient
Average monthly (percent) compliance with daprodustat daily dosing, per subject report. | 120 days
  The average monthly compliance will be calculated from individual subject reported verbal estimates of (percent) compliance with daprodustat daily administration.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Block, MD, Principal Investigator — US Renal Care
Locations (1):
- USRC Kidney Research, Lone Tree, Colorado, United States

IPD SHARING:
Plan to Share IPD: No